CLINICAL TRIAL: NCT00147589
Title: Peds I (Pediatric Eplerenone Development Study I): A Randomized, Double-Blind, Placebo Withdrawal, Parallel Group, Dose-Response Study To Evaluate The Efficacy And Safety Of Eplerenone In The Treatment Of Hypertension In Children
Brief Title: A Study to Evaluate the Efficacy and Safety of Eplerenone in the Treatment of Hypertension in Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6141001
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
To evaluate the efficacy, safety, and toleration of eplerenone in the treatment of children aged 6 to 16 years with high blood pressure. The study will last approximately 10 weeks and about 320 patients will participate.

ELIGIBILITY:
Inclusion Criteria:

* 6-16 years old male and female
* Systolic blood pressure greater than or equal to the 95th percentile for age, gender, and height, measured on at least 3 separate occasions

Exclusion Criteria:

* K/DOQI classification of stages of chronic kidney disease equal to or greater than 3
* Serum or whole blood potassium > 5.5 mEq/L

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320
Dates: Start 2004-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of eplerenone in children

SECONDARY OUTCOMES:
Safety and tolerability of eplerenone in hypertensive children

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (28):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Inglewood, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, Carrboro, North Carolina
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Pittsboro, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Youngstown, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Katy, Texas
- Pfizer Investigational Site, Santo Domingo, DN, Dominican Republic
- India (2):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
- South Africa (7):
  - Pfizer Investigational Site, Capital Park, Gauteng
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Soweto, Gauteng
  - Pfizer Investigational Site, Polokwane, Lipompo Province
  - Pfizer Investigational Site, Parow, Western Cape
  - Pfizer Investigational Site, Cape Town

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141001&StudyName=A+study+to+evaluate+the+efficacy+and+safety+of+Eplerenone+in+the+treatment+of+hypertension+in+children%2E++